CLINICAL TRIAL: NCT06464289
Title: Surgical Stabilisation of Rib Fractures in Non-ventilated Patients: a Retrospective Propensity-matched Analysis Using the Data From the German National Trauma Registry (TraumaRegister of the German Trauma Society (DGU))
Brief Title: Surgical Stabilisation of Rib Fractures in Non-ventilated Patients
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: TraumaRegister® DGU (Unknown)
Responsible Party: Sponsor
Other Study IDs: UKM_UCH_2024_001; 2023-007 (Other: TraumaRegister DGU)
Record Dates: First submitted 2024-05-31; First posted 2024-06-18 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Rib Fractures; Thorax; Fracture
Keywords: surgical stabilisation of rib fractures; non-ventilator-dependent
MeSH Terms: conditions — Rib Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Operative: Patients receiving surgical stabilisation of rib fractures (SSRF) by any operative technique
  Interventions: Procedure: Surgical stabilisation of rib fractures (SSRF); Other: Non-operative management of rib fractures
- Non-operative: Patients not receiving surgical stabilisation of rib fractures (SSRF)
  Interventions: Other: Non-operative management of rib fractures

INTERVENTIONS:
Procedure: Surgical stabilisation of rib fractures (SSRF) — Surgical stabilisation of rib fractures using any fixation technique (including but not limited to plate fixation, intramedullary fixation, wire fixation) via any operative approach (including but not limited to open external approach, minimally invasive approach, thoracoscopic approach, thoracotomy approach).
  Groups: Operative
Other: Non-operative management of rib fractures — Any supportive or specific treatment of rib fractures excluding surgical stabilisation of rib fractures. This includes, but is not limited to analgesia, physiotherapy, non-invasive ventilation, mechanical ventilation, oxygen-supplementation.

SUMMARY:
The aim of the study is to investigate the effect of surgical stabilisation of rib fractures on clinical outcomes in patients that are not dependent on mechanical ventilation at the time of the treatment decision. To this end, data on all eligible patients will be extracted from the TraumaRegister® DGU. Baseline demographics will be analysed using descriptive statistics. Propensity matching will be conducted between the operative cohort (receiving SSRF by any technique) and the conservative cohort (not receiving SSRF). The effect of SSRF on the outcome variables will then be assessed using appropriate statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Rib AIS of ≥ 3
* Initial hospital treatment

Exclusion Criteria:

* Intubated preclinically or in the emergency department
* Glasgow coma scale (GCS) < 9 at the time of the primary survey in the emergency department
* No in-patient hospital management

Ages: 10 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients within the dataset of the TraumaRegister DGU
Sampling Method: Probability Sample
Enrollment: 35974 (Actual)
Dates: Start 2024-04-13 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  Number of patients who died in the hospital and mortality rate up to hospital discharge
Duration of mechanical ventilation | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  The duration in hours a patient spent intubated from the time of hospital admission to the time of initial hospital discharge
Duration of intensive care unit stay. | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  The duration in days a patient spent in the intensive care unit from the time of hospital admission to the time of initial hospital discharge.

SECONDARY OUTCOMES:
Proportion of patients intubated at any time | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  Proportion of patients intubated at any time from time of injury to initial hospital discharge
Duration of hospital stay | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  Duration of the initial hospital stay in days
Rate of single organ failure | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  The Rate of single organ failure from injury to initial hospital discharge
Rate of multiorgan failure | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  The Rate of multiorgan failure from injury to initial hospital discharge
Rate of respiratory failure | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  The Rate of respiratory failure from injury to initial hospital discharge
Rate of sepsis | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  The Rate of sepsis from injury to initial hospital discharge
Clinical outcome | At the time of initial hospital discharge or death, whichever came first, assessed up to 2 month.
  Clinical outcome according to the Glasgow Outcome Scale

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Rosslenbroich, PD Dr. med., Study Director — Department for trauma, hand and reconstructive surgery, University hospital Muenster
Locations (1):
- Department for trauma, hand and reconstructive surgery, University hospital Muenster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huelskamp MD, Duesing H, Lefering R, Raschke MJ, Rosslenbroich S; TraumaRegister DGU. Surgical stabilisation of rib fractures in non-ventilated patients: a retrospective propensity-matched analysis using the data from the trauma registry of the German Trauma Society (TraumaRegister DGUⓇ). Eur J Trauma Emerg Surg. 2025 Jan 24;51(1):55. doi: 10.1007/s00068-024-02756-9. PMID 39856261